CLINICAL TRIAL: NCT01199055
Title: Phase 1b Study of CS-7017 in Combination With Carboplatin/Paclitaxel in Chemotherapy-naïve Subjects With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: CS-7017 in Combination With Carboplatin/Paclitaxel in Subjects With Stage IIIb/IV Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-A108
Record Dates: First submitted 2010-08-30; First posted 2010-09-10 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: PPAR gamma agonist; Tumor; Cancer; Antineoplastic Agent; Respiratory Tract Neoplasms; Carboplatin; Paclitaxel; Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Respiratory Tract Neoplasms | interventions — efatutazone; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-7017+Carboplatin/Paclitaxel (Experimental): Drug: CS-7017 from 0.25 mg twice a day (BID) to 0.50 mg BID for up to 4~6 cycles (1 cycle: 3 weeks)
  Drug: Carboplatin IV, Area under the curve (AUC) of 6 mg/mL*min, once every three weeks for up to 4~6 cycles (1 cycle: 3 weeks)
  Drug: Paclitaxel IV, 200mg/m^2, once every three weeks for up to 4~6 cycles (1 cycle: 3 weeks)
  Interventions: Drug: CS-7017; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: CS-7017 — Drug: CS-7017 from 0.25 mg BID to 0.50 mg BID for up to 4~6 cycles (1 cycle: 3 weeks)
  Other Names: CS7017
Drug: Carboplatin — Drug: Carboplatin IV, AUC of 6 mg/mL*min, once every three weeks for up to 4~6 cycles (1 cycle: 3 weeks)
  Other Names: Paraplatin
Drug: Paclitaxel — Drug: Paclitaxel IV, 200mg/m^2, once every three weeks for up to 4~6 cycles (1 cycle: 3 weeks)
  Other Names: Taxol

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of CS-7017 administered orally twice a day in combination with carboplatin and paclitaxel, and to assess the pharmacokinetics of CS-7017 in combination with carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable locally advanced or metastatic (stage IIIb or IV) non-small cell lung cancer (NSCLC)
* No prior systemic therapy for NSCLC
* Male or female ≥ 18 years of age
* Anticipation of more than 3 months survival
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or radiation therapy during the study
* Remaining influence of previous therapies such as radiotherapy, surgery, immunotherapy within 4 weeks prior to start of study treatment
* History of any of the following events within 6 months prior to start of study treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class ≥I congestive heart failure (CHF), cerebrovascular accident or cerebral infarction, pulmonary embolism, deep vein thrombosis, or other clinically significant thromboembolic event; clinically significant pulmonary disease (eg, severe chronic-obstructive pulmonary disease (COPD) or asthma)
* Severe edema, ascites fluid, pericardial or pleural effusion or pericardial involvement with the tumor within 6 months prior to start of study treatment, or which require steroid therapy/ diuretic therapy
* Subjects with brain metastasis (defined as untreated, symptomatic or requiring steroids or anticonvulsant medications to control associated symptoms)
* Subjects with clinically significant active infection which requires antibiotic therapy, or who are hepatitis B surface antigen (HBs)- or hepatitis C virus (HCV)- or human immunodeficiency virus (HIV)- positive and receiving antiretroviral therapy
* Subjects with malabsorption syndrome, chronic diarrhea (lasting over 4 weeks), inflammatory bowel disease, or partial bowel obstruction
* Diabetes mellitus requiring insulin, or a history of poor serum glucose control with the use of non-insulin diabetes medications
* Treatment with thiazolidinediones (TZDs) within 4 weeks prior to start of study treatment
* History of a second malignancy, with the exception of in situ cervical cancer or adequately treated basal cell or squamous cell carcinoma of the skin
* Poorly-controlled blood pressure as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 participants were screened for eligibility. Of the 18 participants who were screened, 16 participants who met all inclusion criteria and no exclusion criteria were enrolled from 17 March 2010 to 15 April 2011 at 1 site in South Korea. All 16 participants received treatment.
Pre-assignment Details: This dose-escalating study included an initial and additional portion. Participants received CS-7017 combination treatment with carboplatin & paclitaxel (starting dose 0.25 mg twice daily [BID] in the initial portion). In the additional portion, the CS-7017 dose was determined (0.50 mg BID) based on the initial portion.
Groups:
- CS-7017 0.25 mg BID; Initial Portion: Participants who received 0.25 mg twice daily (BID) CS-7017 combination treatment administered orally. Paclitaxel was administered intravenously at a dose of 200 mg/m^2 over 3 hours immediately after administration of CS-7017. Carboplatin was administered intravenously. The dose of the carboplatin was calculate using Calvert formula and target area under the plasma concentration-time curve (AUC) of 6 mg/mL*min.
- CS-7017 0.50 mg BID; Initial Portion: Participants who received 0.50 mg twice daily (BID) CS-7017 combination treatment administered orally. Paclitaxel was administered intravenously at a dose of 200 mg/m^2 over 3 hours immediately after administration of CS-7017. Carboplatin was administered intravenously. The dose of the carboplatin was calculate using Calvert formula and target area under the plasma concentration-time curve (AUC) of 6 mg/mL*min.
- CS-7017 0.50 mg BID; Additional Portion: Participants who received 0.5 mg twice daily (BID) CS-7017 combination treatment administered orally. Paclitaxel was administered intravenously at a dose of 200 mg/m^2 over 3 hours immediately after administration of CS-7017. Carboplatin was administered intravenously. The dose of the carboplatin was calculate using Calvert formula and target area under the plasma concentration-time curve (AUC) of 6 mg/mL*min.
  Cycle 1, Day 1: Carboplatin and paclitaxel only
  Cycle 1, Day 3: CS-7017 at the dose selected in initial portion
  Subsequent cycles: CS-7017 with carboplatin and paclitaxel
Period: Overall Study
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Started | 3 | 4 | 9
Completed | 1 | 1 | 5
Not Completed | 2 | 3 | 4
Not completed — Death | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Progressive disease | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | Total
Number analyzed (Participants) | 3 | 4 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 10
  >=65 years | 1 | 2 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.29) | 62.3 (5.91) | 58.9 (9.98) | 59.9 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 5
  Male | 2 | 4 | 5 | 11
Region of Enrollment [Number; unit: participants]
  South Korea | 3 | 4 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve of Geometric Means of Serum Free Form of CS-7017 (R-150033) After Administration of CS-7017 and Carboplatin/Paclitaxel in Participants With Stage IIIb/IV Non-small Cell Lung Cancer
Description: The area under the concentration versus time curve during dosing interval (AUCtau) and up to the last quantifiable time (AUClast) of geometric means of CS-7017 are reported at selected cycles (C) and days (D).
Time Frame: Initial C1D1, C2D22 and additional C1D3, C2D22 predose, 0.5, 1, 2, 3, 4, 6 and 10h; initial and additional D8 predose; additional D1 predose and 3h; initial and additional D15 predose and 1-3h; C3D43 and C4D64 any time, except additional C3D43 predose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Number analyzed (Participants) | 3 | 4 | 9
ng*h/mL
  Cycle 1, Week 1: AUCtau: number analyzed (Participants) | 3 | 2 | 3
  Cycle 1, Week 1: AUCtau | 70.66 (54.11) | 209.33 (131.40) | 203.99 (91.34)
  Cycle 1, Week 1: AUClast | 49.57 (36.86) | 87.23 (85.69) | 81.54 (66.01)
  Cycle 2, Week 4: AUCtau: number analyzed (Participants) | 3 | 3 | 4
  Cycle 2, Week 4: AUCtau | 132.47 (25.49) | 345.56 (156.29) | 400.89 (212.22)
  Cycle 2, Week 4: AUClast: number analyzed (Participants) | 3 | 3 | 5
  Cycle 2, Week 4: AUClast | 95.94 (15.84) | 240.61 (107.09) | 268.00 (134.40)

2. Primary Outcome: Pharmacokinetic Parameter Observed Serum Concentration (Cmax) of Geometric Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 and Carboplatin/Paclitaxel in Participants With Stage IIIb/IV Non-small Cell Lung Cancer
Description: The maximum serum concentration (including at steady state (ss) of CS-7017 are reported at selected cycles (C) and days (D).
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Number analyzed (Participants) | 3 | 4 | 9
ng/mL
  Cycle 1, Week 1: Cmax | 8.90 (7.01) | 15.98 (16.77) | 14.54 (9.75)
  Cycle 2, Week 4: Cmax,ss: number analyzed (Participants) | 3 | 3 | 5
  Cycle 2, Week 4: Cmax,ss | 13.63 (1.77) | 33.83 (15.42) | 39.58 (18.63)

3. Primary Outcome: Pharmacokinetic Parameter Time of Maximum Plasma Concentration (Tmax) of Geometric Means of Serum Free Form of CS-7017 (R-150033) Following Administration of CS-7017 and Carboplatin/Paclitaxel in Participants With Stage IIIb/IV Non-small Cell Lung Cancer
Description: The time of maximum plasma concentration (including at steady state (ss) of CS-7017 are reported at selected cycles (C) and days (D).
Time Frame: as for outcome 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: h
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Number analyzed (Participants) | 3 | 3 | 9
h
  Cycle 1, Week 1: Tmax | 3.90 [1.98 to 3.95] | 3.00 [2.92 to 6.05] | 5.95 [2.00 to 8.10]
  Cycle 2, Week 4: Tmax,ss: number analyzed (Participants) | 3 | 3 | 5
  Cycle 2, Week 4: Tmax,ss | 3.17 [3.02 to 4.08] | 3.98 [2.90 to 4.12] | 3.88 [1.95 to 6.02]

4. Primary Outcome: Treatment-Emergent Adverse Events Occurring in Participants in Any Treatment Group During Cycle 1 Following Administration of CS-7017 and Carboplatin/Paclitaxel in Participants With Stage IIIb/IV Non-small Cell Lung Cancer
Description: Treatment-emergent adverse events (TEAEs) are defined as those adverse events that occur, having been absent before the study, or worsen in severity after the initiation of study drug.
Time Frame: Baseline to end of Cycle 1, with each treatment cycle being 3 weeks
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Number analyzed (Participants) | 3 | 4 | 9
Participants
  At least one TEAE | 3 | 4 | 9
  Blood and lymphatic system disorders | 3 | 2 | 8
  Neutropenia | 3 | 2 | 7
  Anaemia | 0 | 0 | 5
  Metabolism and Nutrition Disorders | 0 | 2 | 6
  Decreased appetite | 0 | 1 | 6
  Nervous System Disorders | 1 | 1 | 4
  Neuropathy peripheral | 0 | 1 | 4
  Respiratory, Thoracic and Mediastinal Disorders | 1 | 0 | 4
  Pleural effusion | 0 | 0 | 4
  Gastrointestinal Disorders | 2 | 1 | 6
  Nausea | 2 | 1 | 1
  Skin and Subcutaneous Tissue Disorders | 2 | 2 | 8
  Alopecia | 2 | 1 | 8
  Pruritus | 0 | 2 | 1
  Musculoskeletal and Connective Tissue Disorders | 3 | 2 | 7
  Myalgia | 2 | 0 | 6
  Athralgia | 1 | 2 | 0
  General Disorders & Administration Site Conditions | 3 | 1 | 5
  Fatigue | 3 | 0 | 1
  Investigations | 0 | 2 | 8
  Weight increased | 0 | 2 | 7

5. Secondary Outcome: Best Overall Response and Objective Response Rate Following Administration of CS-7017 in Combination With Carboplatin/Paclitaxel in Chemotherapy-naïve Subjects With Metastatic or Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Description: The best overall response is the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], stable disease [SD], and progressive disease [PD]) among all overall responses from the start of treatment until the participant withdraws from the study. Participants who did not have a tumor assessment, the best overall response is Not Evaluable (NE). The response rate was defined as the proportion of participants with a best overall response of CR or PR, ie, [confirmed and unconfirmed, (CR + PR) / number of participants]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, CR was defined as the disappearance of all target lesions, PR was defined as ≥30% decrease in the sum of diameters of target lesions, PD was defined as ≥20 increase in the smallest sum of diameters, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline up to Week 18 postdose
Population: Best overall response and objective response rate were assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- CS71017 0.5 mg BID; Initial and Additional Portion: All participants who received 0.5 mg twice daily CS-7017 in combination with carboplatin and paclitaxel during either the initial or additional portion.
- Overall: All participants who received CS-7017 in combination with carboplatin and paclitaxel.
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion | CS71017 0.5 mg BID; Initial and Additional Portion | Overall
Number analyzed (Participants) | 3 | 3 | 8 | 11 | 14
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 2 | 4 | 6 | 6
  Stable disease (SD) | 1 | 0 | 2 | 2 | 3
  Progressive disease (PD) | 2 | 1 | 2 | 3 | 5
  Not evaluable (NE) | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0
  Response rate (CR + PR) | 0 | 2 | 4 | 6 | 6

6. Secondary Outcome: CS-7017-Related Treatment-Emergent Adverse Events Occurring in Participants in Any Treatment Group After Administration of CS-7017 and Carboplatin/Paclitaxel in Chemotherapy-naïve Participants With Stage IIIb/IV Non-small Cell Lung Cancer
Description: Treatment-emergent adverse events (TEAEs) are defined as those adverse events that occur, having been absent before the study, or worsen in severity after the initiation of study drug. CS-7017-related TEAEs are those TEAEs that are related to CS-7017 in the relationship.
Time Frame: Baseline to 30 days after last dose, up to approximately 1 year
Population: CS-7017-related TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
Number analyzed (Participants) | 3 | 4 | 9
Participants
  At least one CS-7017-related TEAE | 2 | 3 | 8
  Respiratory, Thoracic and Mediastinal Disorders | 0 | 1 | 4
  Pleural effusion | 0 | 1 | 4
  General Disorders & Administration Site Conditions | 1 | 2 | 7
  Face oedema | 1 | 2 | 4
  Oedema peripheral | 0 | 2 | 3
  Investigations | 1 | 3 | 8
  Weight increased | 1 | 3 | 8

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event data were collected from baseline to 30 days after last dose, up to approximately 1 year.
Description: Adverse events were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within the 30 days after the last dose of the study drug.
Arm/Group | CS-7017 0.25 mg BID; Initial Portion | CS-7017 0.50 mg BID; Initial Portion | CS-7017 0.50 mg BID; Additional Portion
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 6/9
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.25 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Initial Portion (N=4) | CS-7017 0.50 mg BID; Additional Portion (N=9)
Pyrexia (General disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Weight increased (Investigations) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.25 mg BID; Initial Portion (N=3) | CS-7017 0.50 mg BID; Initial Portion (N=4) | CS-7017 0.50 mg BID; Additional Portion (N=9)
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 9
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 7
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 9
Dizziness (Nervous system disorders) | 3 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 8
Constipation (Gastrointestinal disorders) | 1 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6
Athralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Asthenia (General disorders) | 2 | 2 | 7
Fatigue (General disorders) | 3 | 1 | 4
Face oedema (General disorders) | 1 | 2 | 4
Oedema peripheral (General disorders) | 0 | 2 | 3
Weight increased (Investigations) | 1 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No